CLINICAL TRIAL: NCT07295041
Title: Allogenic Bone Blocks and Particulate Graft for Horizontal Bone Augmentation in the Posterior Mandible: a Randomized Controlled Trial
Brief Title: GBR Versus Allogenic Bone Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Algirdas Puisys, DDS, PhD (Network)
Responsible Party: Sponsor-Investigator, Algirdas Puisys, DDS, PhD, DDS, PhD, Vilniaus Implantologijos Centro (VIC) Klinika
Organization: Vilniaus Implantologijos Centro (VIC) Klinika (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEC-LSMU(R)-51
Record Dates: First submitted 2025-11-24; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Alveolar Bone Grafting; Implant Placement
Keywords: bone block, GBR; guided bone regeneration; allogenic graft; bone particulate; allogenic bone block; allogenic bone particulate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- allogenic bone blocks (Active Comparator): Patients in this group received allogenic bone blocks for the primary bone augmentation procedure.
  Interventions: Procedure: allogenic bone blocks
- allogenic cancellous bone granules (Active Comparator): Patients in this group received allogenic cancellous bone granules for the primary bone augmentation procedure.
  Interventions: Procedure: allogenic cancellous bone granules

INTERVENTIONS:
Procedure: allogenic bone blocks — An allogenic bone blocks were used for the primary bone augmentation procedure.
  Arms: allogenic bone blocks
Procedure: allogenic cancellous bone granules — allogenic cancellous bone granules were used for the primary bone augmentation procedure.
  Arms: allogenic cancellous bone granules

SUMMARY:
This study aimed to compare two different methods used to augment bone in the posterior lower jaw prior to implant placement in patients with insufficient bone width. Eligible patients were included in the study and received a horizontal bone augmentation with one of two methods, which differed in the materials used for the bone augmentation. The group allocation was randomised. After 6 months of healing following parameters were assessed: histological evaluation, survival of the bone graft, the need for further bone augmentation at the time of implant placement, changes in soft tissue characteristics, radiologically and clinically assessed changes in bone width.

DETAILED DESCRIPTION:
Objective: The objective of this study is to compare the histological, clinical, and radiographic outcomes of particulate bone substitutes versus allogenic bone block grafts for primary bone augmentation in the posterior mandible.

Materials and Methods: This randomised controlled clinical trial included adult patients in need for a staged bone augmentation prior to implant placement in the posterior mandible. Patients were randomly assigned to one of two treatments groups. Patients allocated in the BBL group received allogenic bone blocks, whereas patients in the GBR group received allogenic bone granules for the primary bone augmentation. In both groups grafting materials were covered with a resorbable collagen membrane, which was fixated with non-resorbable fixation pins. The primary outcome of this study was defined as the composition of the histological samples at least 6 months after the primary bone augmentation. Secondary outcomes included graft survival rates, the need for further augementation procedures at time of implant placement, soft tissue measurements and radiographically and clinically analyzed changes in bone width and radiographically analyzed changes in bone volume. These outcomes were measured at baseline (prior to bone augmentation surgery) and at the follow-up (at least 6 months after bone augmentation).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Insufficient bone width in posterior mandible requiring staged bone augmentation prior to implant placement
* Minimum of 1 mm bone width available
* Willing to provide signed informed consent

Exclusion Criteria:

* Pregnant or lactating
* Known or suspected incompliance
* Patients smoking more than 10 cigarettes per day
* Systemic diseases or medications affecting bone metabolism (such as osteoporosis, intake of bisphosphonates)
* Active periodontal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Histological composition | 6 months
  Histological samples were obtained at the time of reentry for implant placement at least 6 months after the primary bone augmentation procedure. Sample analysis included the measurement of the total sample area, the area of identified bone, biomaterial and soft tissue per sample. Furthermore, the percentage of bone, biomaterial and soft tissue per sample was calculated.

SECONDARY OUTCOMES:
Need for further augmentation procedures at the time of implant placement | 6 months
  The need for further soft and hard tissue augmentation procedures at the time of implant placement was evaluated at the time of implant placement.
Keratinized tissue height | Baseline and 6 months
  keratinized tissue height measured with a periodontal probe at baseline and follow-up.
Vertical soft tissue thickness | Baseline and 6 months
  the vertical soft tissue thickness measured with a periodontal probe at baseline and follow-up.
Clinically measured bone width | Baseline and 6 months
  the bucco-oral bone width measured with a periodontal probe at baseline and follow-up.
Radiologically measured bone width | Baseline and 6 months
  Bucco-oral bone width in the augmented region was measured on baseline and follow-up CBCTs.
Changes in bone volume | Baseline and 6 months
  CBCT images prior to bone augmentation and after the healing period were superimposed. The changes in bone volume in the augmented area were measured.

CONTACTS AND LOCATIONS:
Locations (1):
- VIC Klinika, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No